CLINICAL TRIAL: NCT02335840
Title: Influence of Different Doses of Coffee in the Blood Pressure Response Post-exercise
Brief Title: Doses of Coffee and Blood Pressure Response Post-exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Alesandra Araújo de Souza, Master Student, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 21/2011
Record Dates: First submitted 2014-12-23; First posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Post-Exercise Hypotension; Hypertension
MeSH Terms: conditions — Post-Exercise Hypotension; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- One dose of coffee (Experimental): Ingestion of one dose of 150 ml of coffee (144 mg of caffeine) ingested 10 minutes post-exercise (denominated CAF-1)
  Interventions: Other: CAF-1
- Two doses of coffee (Experimental): Ingestion of two doses of 150 ml of coffee (144 mg of caffeine) ingested 10 and 20 minutes post-exercise (denominated CAF-2)
  Interventions: Other: CAF-2
- Three doses of coffee (Experimental): Ingestion of three doses of 150 ml of coffee (144 mg of caffeine) ingested 10, 20 and 30minutes post-exercise (denominated CAF-3)
  Interventions: Other: CAF-3
- Three doses of decaffeinated coffee (Experimental): Ingestion of three doses of 150 ml of decaffeinated coffee (144 mg of caffeine) ingested 10, 20 and 30 minutes post-exercise (denominated DESC)
  Interventions: Other: DESC

INTERVENTIONS:
Other: CAF-1 — In this intervention the volunteers ingested one dose of caffeinated coffee containing 144 mg of caffeine
  Arms: One dose of coffee
Other: CAF-2 — In this intervention the volunteers ingested two doses of caffeinated coffee containing 288 mg of caffeine
  Arms: Two doses of coffee
Other: CAF-3 — In this intervention the volunteers ingested three doses of caffeinated coffee containing 432mg of caffeine
  Arms: Three doses of coffee
Other: DESC — In this intervention the volunteers ingested one dose of decaffeinated coffee containing 108 mg of caffeine
  Arms: Three doses of decaffeinated coffee

SUMMARY:
Introduction: reduction of blood pressure after physical exercise is called post exercise hypotension (PEH). However, previous studies demonstrate that ingestion of caffeine equivalent to three tea-cup of coffee abolishes this phenomenon. Objective: evaluate the influence of different doses of coffee in PEH. Methods: eleven hypertensive performed four experimental sessions of aerobic exercise in cycle ergometer (40 minutes of duration, intensity between 60% and 80% of maximum heart rate) succeeds for the ingestion of one (CAF-1), two (CAF-2), three (CAF-3) doses of caffeinated coffee (144 mg/dose), or three doses of decaffeinated coffee (DESC). Blood pressure was measured in rest and during 120 minutes of recovery post exercise, each 10 minutes.

DETAILED DESCRIPTION:
Volunteers: participated 12 volunteers diagnosed as hypertensive, both gender (three men), 40 to 55 years old, overweight and practitioners of aerobic exercise (walk) at least three months. They were treated with anti-hypertensive medication of class beta-adrenergic receptor blockers, thiazides and enzyme convertor of angiotensin inhibitors, and showing systolic and diastolic pressoric values controlled and habituated to coffee consumption. Would be excluded from the study volunteers who presented migraine or other withdrawal symptoms due to a washout to be carried out for coffee and other caffeinated foods. The volunteers participated of this study for average one month. This study was previously approved by Ethic Committee in Search with Humans at Hospital Lauro Wanderley, at Federal University of Paraiba, under protocol 21/2011. All volunteers was previously clarified about the experimental procedures, and they signed the written informed consent according resolution 466/12 at Health National Council (Brazil).

Design of Study: the study was experimental, randomized and double-blind. Before the experimental sessions the volunteers were instructed to avoid caffeinated foods during 48 hours. They performed four experimental sessions with the practice of aerobic exercise, succeed for the ingestion of caffeinated or decaffeinated coffee, according to following protocols: 1) one dose of 150 ml of coffee (144 mg of caffeine) ingested 10 minutes post-exercise (CAF-1); 2- two doses of 150 ml of coffee (2x144 mg of caffeine) ingested 10 and 20 minutes post-exercise (CAF-2); three doses of 150ml of coffee (3x 144 mg of caffeine) ingested 10, 20 and 30 minutes post-exercise (CAF-3); 4- three doses of 150 ml of decaffeinated coffee (108 mg of caffeine) ingested 10, 20 and 30 minutes post-exercise (DESC). The order of realization experimental sessions was determined randomly through the site www.randomizer.org. They remained seated during 120 minutes after exercise. Blood pressure was evaluated in rest, and during 120 minutes of post-exercise recovery, each 10 minutes.

Preparation and Ingestion of coffee: was utilized one caffeinated and decaffeinated coffee (São Braz, Cabedelo, Brazil) with one same serial number. Caffeinated and decaffeinated coffee had 1,2% and 0,3% of caffeine, respectively, in your composition. The method adopted to the preparation of caffeinated or decaffeinated coffee was previously utilized for Nóbrega et al. (15). Were prepared with addition of 40g coffee powder to each 500 ml of heated water during five minutes, limited by beginning of boil. Thus, the volume of 500 ml of coffee had one concentration of 480 mg of caffeine. Considering each tea-cup ingested had one volume of 150 ml, so one, two and three tea-cups with coffee had respectively 144 mg, 288 mg and 432 mg of caffeine. Three tea-cups of decaffeinated coffee were 108 mg of caffeine. The doses of caffeinated or decaffeinated coffee were sweetened with sugar (Alegre, Mamanguape, Brazil). The coffee was strained with filters paper (Mellita®, Minden, Alemanha). To ensure the accuracy of volume intake by volunteers at all time was utilized one dosing tea-cup previously calibrated to volume of one tea-cup (150 ml). The intake coffee was performed on first 30 minutes of period recovery, each 10 minutes. During moment of ingestion, volunteers stay seated and was stipulated a deadline of five minutes to intake the coffee.

Protocol of Physical Exercise: volunteers performed four experimental sessions with aerobic exercise on a stationary bicycle (Perform V3, Movement®, Pompeia, Sao Paulo), lasting 40 minutes, intensity between 60 and 80% of maximum heart rate (MHR). To estimate of MHR was utilized the equation proposed by Bruce et al. (16). To the prescription of target zone for exercise was adopted the protocol proposed by Karvonen et al. (17). The heart rate of rest and during the exercise was evaluated utilizing by cardiofrequencymeter (RS800CX, Polar Electro® Oy, Kempele, Finland)

Measures of Blood Pressure: after the volunteers arrived on laboratory, they were oriented to stay in rest seated during 10 minutes to measures of blood pressure on end of this period. Others measures were realized during the 120 minutes of post-exercise recovery, each 10minutes. The first 30 minutes of post-exercise recovery the measures were always performed one minute before coffee administration. The blood pressure was measured by auscultatory method, following the protocol proposed by VI Brazilian Guidelines of Arterial Hypertension (18). For this, was utilized one sphygmomanometer (Missouri, Embu, Brasil), previously calibrated against one mercury column and one stethoscope (Missouri, Embu, Brasil).

Statistical Analysis: all the data are presented as mean±standard-error of mean. All variables were tested for normal distribution using Shapiro-Wilk and Levene tests. For the comparisons of age, body mass index, heart rate of rest, systolic and diastolic blood pressure of rest between the experimental sessions was utilized one-way ANOVA. For the comparisons of systolic and diastolic post-exercise between the experimental sessions of study was realized two-way ANOVA plus Bonferroni test post hoc. P value small than 0,05 was considered statically significant.

ELIGIBILITY:
Inclusion Criteria:

* Were included subjects of both gender (three men), 40 to 55 years old, overweight and practitioners of aerobic exercise (walk) at least three months. They were treated with anti-hypertensive medication of class beta-adrenergic receptor blockers, thiazides and enzyme convertor of angiotensin inhibitors, and showing systolic and diastolic values controlled and habituated to coffee consumption.

Exclusion Criteria:

* Would be excluded from the study volunteers who presented migraine or other withdrawal symptoms due to a washout to be carried out for coffee and other caffeinated foods.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure. The measures were evaluated for delta (difference between the values obtained in the period of recovery and baseline) | The systolic and diastolic blood pressure were measured in CAF-1, CAF-2, CAF-3 and DESC after the baseline and during 120 minutes post-exercise each 10 minutes. Thus, were realized 13 measures of blood pressure in each experimental session.
  The sessions CAF-1, CAF-2, CAF-3 and DESC were realized with interval of 72 hours between them, thus, each volunteer devoted an average 20 days to the study.